CLINICAL TRIAL: NCT01704898
Title: Comparative Bioavailability Study of Two Efavirenz 600 mg Formulations in Healthy Volunteers.
Brief Title: Efavirenz Comparative Bioavailability
Acronym: efv600
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Center for Clinical Pharmacology Research Bdbeq S.A. (Other)
Collaborators: University of the Republic, Uruguay (Other)
Responsible Party: Principal Investigator, Francisco E. Estevez-Carrizo, M.D., Chief Medical Officer, Center for Clinical Pharmacology Research Bdbeq S.A.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: bdbeq-efv600/icuvita-020
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: efavirenz; bioequivalence; fasting; healthy volunteers
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Efavirenz 600 Test-Stocrin 600 Reference (Other): Efavirenz 600 mg will be randomly assigned.
  Interventions: Drug: Efavirenz 600 Test-Stocrin 600 Reference
- Stocrin 600 Reference-Efavirenz 600 Test (Other): Stocrin 600 mg will be randomly assigned.
  Interventions: Drug: Stocrin 600 Reference-Efavirenz 600 Test

INTERVENTIONS:
Drug: Efavirenz 600 Test-Stocrin 600 Reference
  Arms: Efavirenz 600 Test-Stocrin 600 Reference
Drug: Stocrin 600 Reference-Efavirenz 600 Test
  Arms: Stocrin 600 Reference-Efavirenz 600 Test

SUMMARY:
The primary objective of this study is to determine the average bioequivalence of a generic efavirenz 600 mg tablet (test formulation)compared with Stocrin(R) 600 mg tablets (Reference formulation).The study is designed as an open label, randomized, crossover, 2-treatments, 2-period, 2-sequence, single dose pharmacokinetic study conducted in healthy volunteers. Subjects will be randomized to receive generic efavirenz 600 (Test formulation) or Stocrin(R) 600 tablets (Reference formulation)on study day 1 (period 1). Subjects will undergo a 24 hour intensive pharmacokinetic evaluation after ingesting a single dose of either the Test or Reference formulation. Subjects will provide additional pharmacokinetic samples 36, 48, 72, 120 and 192 hours postdose, respectively. Subjects will complete a wash out period from day 8 to day 28 during wich no study drug will be ingested. On day 29 subjects will ingest either the Test or the Reference formulation (opposite to the formulation received on period 1). All subjects undergo another 24 hour intensive pharmacokinetic evaluation and pharmacokinetics samples on days 36, 48, 72, 120, 192 pos dose, respectively. Adverse events and and concomitant medication will be documented throughout the study.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the average bioequivalence of generic efavirenz 600 mg tablet (test formulation)compared with Stocrin(R) 600 mg tablets (Reference formulation).The study is designed as an open label, randomized, crossover, 2-treatments, 2-period, 2-sequence, single dose pharmacokinetic study conducted in healthy volunteers.

Subjects will be randomized to receive generic efavirenz 600 (Test formulation) or Stocrin(R) 600 tablets (Reference formulation)on study day 1 (period 1), then they will undergo a 24 hour intensive pharmacokinetic evaluation after ingesting a single dose of either the Test or Reference formulation. Additional pharmacokinetic samples 36, 48, 72, 120 and 192 hours postdose will be drawn.

Subjects will complete a wash out period form day 8 to day 28 during which no study drug will be ingested. On day 29 (period 2) they will ingest either the Test or the Reference formulation (opposite to the formulation received on period 1). All subjects undergo another 24 hour intensive pharmacokinetic evaluation and pharmacokinetics samples on days 36, 48, 72, 120, 192 pos-dose, respectively, will be drawn. Adverse events and concomitant medication will be documented throughout the study.

The sample size is 28 and is based on a 15% dropout rate (due to lost to follow-up, treatment discontinuation, etc.) Since the investigators are expecting four subjects not to complete the study,24 evaluable subjects are finally expected. If the discontinuation rate is greater than 15%, the investigators will continue to enroll until they get 24 evaluable subjects.

The primary endpoint is to determine average bioequivalence for Test and Reference formulation of efavirenz according to the FDA guidance on bioequivalence testing. The ratio of the Test to Reference formulation mean for efavirenz AUC0-192, AUC0-inf and Cmax and the 90% confidence interval around each mean ratio will be determined. Average bioequivalence will be met if 90% confidence interval around de AUC and Cmax mean ratios for efavirenz falls within the FDA's predefined limits of 0.80 to 1.25.

Safety will be evaluated by administering a questionnaire to the subjects during the study . This questionnaire will list the most frequent adverse effects already described for the innovator (Stocrin(R)). Safety will also be evaluated from vital signs recordings, lab tests out of the limits fixed in the study protocol and Psychiatric Evaluations during screening, in the wash out period and 15 days after the last administration of the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Male,
* Caucasians
* Age >=18 and <=50,
* BMI>18 and BMI<30 kg/m2
* HIV-1 negative, B Hepatitis negative, C Hepatitis negative.
* Able to give consent,
* Non/light-smoking,
* Lab screening and EKG within the limits stipulated in the protocol.
* Healthy as determine by medical examination.

Exclusion Criteria:

* Subjects with any current or past history of psychiatric disorder.
* Subjects receiving any prescription or over-the-counter product.
* Subjects using any form of recreational drug.
* Subjects who has eaten grapefruit or drunk grapefruit juice during the last 15 days before administration of study drug.
* Subjects who had had xanthine containing beverages (mate, coffee, tea, chocolate, etc.) during 48 ours previous to study drug administration.
* Subjects with history of hepatic disease, renal disease, GI diseases, chronic infectious disease, heart disease, lung disease, neurologic disease, endocrine disease, etc.
* Subjects suffering any acute disease at screening or check-in.
* Alanine S. Transaminase(AST)/Alanine L. Transaminase(ALT) > 3 times upper limit of normal (ULN).
* Bilirubin > 2.5 times ULN.
* Amylase > 2 times ULN.
* Absolute Neutrophil Count <1000/mL.
* Hgb < 9.0 g/dl.
* Platelets > 50.000 cell/mm3,
* Serum Creatinine > 2.5 mg/dl

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve for efavirenz (AUC0-192) | 0 to 192 h
  The area under the concentration-time curve (AUC0-192) for efavirenz in a time frame of 8 days.
Maximum Concentration for efavirenz (Cmax) | 0 to 192 h
  The maximum concentration taken form the curve concentration vs. time for efavirenz.
Area Under the Curve 0 to infinity for efavirenz (AUC0-inf) | 0 to infinity
  Area under the concentration-time curve from time 0 to infinity for efavirenz.

SECONDARY OUTCOMES:
Time to the Cmax for efavirenz (tmax) | 0 to 192 h
  It is the time elapsed from 0 time to the Cmax time for efavirenz

OTHER OUTCOMES:
First order elimination rate constant for efavirenz (Ke) | 0 to 192 h
  It is the firs order efavirenz elimination rate constant, calculated from the final elimination phase of the curve concentration vs. time.
Elimination Half Life (T1/2e) | 0-92 h
  This outcome measures the rate of drug elimination form the body.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco E. Estevez, M.D., Principal Investigator — Center for Clinical Pharmacology Research Bdbeq S.A.
Locations (1):
- Center for Cllinical Pharmacology Research-Bdbeq S.A., Montevideo, Montevideo Department, Uruguay

REFERENCES:
- [Background] Kaul S, Ji P, Lu M, Nguyen KL, Shangguan T, Grasela D. Bioavailability in healthy adults of efavirenz capsule contents mixed with a small amount of food. Am J Health Syst Pharm. 2010 Feb 1;67(3):217-22. doi: 10.2146/ajhp090327. PMID 20101064
- [Background] Mathias AA, Hinkle J, Menning M, Hui J, Kaul S, Kearney BP; Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate Single-Tablet Regimen Development Team. Bioequivalence of efavirenz/emtricitabine/tenofovir disoproxil fumarate single-tablet regimen. J Acquir Immune Defic Syndr. 2007 Oct 1;46(2):167-73. doi: 10.1097/QAI.0b013e3181427835. PMID 17667331
- [Background] Frampton JE, Croom KF. Efavirenz/emtricitabine/tenofovir disoproxil fumarate: triple combination tablet. Drugs. 2006;66(11):1501-12; discussion 1513-4. doi: 10.2165/00003495-200666110-00012. PMID 16906786
- [Background] Marier JF, Morin I, Al-Numani D, Stiles M, Morelli G, Tippabhotla SK, Vijan T, Singla AK, Garg M, Di Marco M, Monif T. Comparative bioavailability of a generic capsule formulation of the reverse transcriptase inhibitor efavirenz and the innovator product. Int J Clin Pharmacol Ther. 2006 Apr;44(4):180-4. doi: 10.5414/cpp44180. PMID 16625987